CLINICAL TRIAL: NCT02900209
Title: Responses of the Immune System to Influenza Vaccination in Phenotypes of Chronic Obstructive Pulmonary Disease
Brief Title: Influenza Vaccination and COPD Phenotypes
Status: Completed | Type: Observational
Sponsor: University of Lincoln (Other)
Collaborators: University of Kent (Other); NHS Lincolnshire West Clinical Commissioning Group (Other); NHS South Lincolnshire Clinical Commissioning Group (Other)
Responsible Party: Principal Investigator, Arwel Jones, Research Fellow, University of Lincoln
Other Study IDs: CoSREC192
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Influenza; Exacerbations
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood samples will be collected in K3EDTA and serum vacutainer tubes. Saliva samples will be obtained while participant is seated with the head tilted slightly forward and passively dribbling into a pre-weighed sterile tube (keeping orofacial movement to a minimum).
  Whole blood samples will be used on the day of collection and analysed before being appropriately disposed of on the same day. Blood samples will be centrifuged with plasma and serum frozen at -80c for later analysis. Saliva samples will also be centrifuged with supernatant frozen at -80c for later analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- COPD frequent exacerbators: Aged 65-85 years with a diagnosis of COPD according to Global Initiative for Chronic Obstructive Lung Disease criteria (post bronchodilator FEV1/FVC ratio <0.70). Moderate to severe airflow limitation (FEV1 30-80% predicted). Patients have experienced 2 or more exacerbations requiring oral steroids/antibiotics treatment and/or hospitalisation in the previous 12 months.
  Interventions: Other: Influenza Vaccination
- COPD infrequent exacerbators: Aged 65-85 years with a diagnosis of COPD according to Global Initiative for Chronic Obstructive Lung Disease criteria (post bronchodilator FEV1/FVC ratio <0.70). Moderate to severe airflow limitation (FEV1 30-80% predicted). Patients have experienced no more than 1 course of oral steroids/antibiotics and none exacerbations requiring hospital admission in the previous 12 months.
  Interventions: Other: Influenza Vaccination
- Healthy controls: Aged 65-85 years and do not have any symptoms of lung disease and have normal spirometry.
  Interventions: Other: Influenza Vaccination

INTERVENTIONS:
Other: Influenza Vaccination

SUMMARY:
The aim of this study is to determine responses of the immune system to the annual flu vaccination in people with COPD who experience frequent or infrequent exacerbations and healthy participants. We will collect blood and saliva immediately before and one month after flu vaccination at GP surgeries in the Autumn/Winter period. By measuring how quickly antibodies (that provide protection against infection) develop in the blood after vaccination we can provide important new information to help confirm whether those prone to COPD flare ups have weaker immune systems.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 65-85 years with a diagnosis of COPD (according to Global Initiative for Chronic Obstructive Lung Disease criteria: post bronchodilator FEV1/FVC ratio <0.70) and moderate to severe airflow limitation (FEV1 30-80% predicted) who opt to receive the annual influenza vaccine.

We will also include healthy participants aged 65-85 years without symptoms of lung disease who opt to receive the annual influenza vaccine.

Exclusion Criteria:

* Unable/unwilling to provide informed consent
* Any history of allergies, suspected hypersensitivity and/or contraindication to vaccines (e.g egg protein allergy)
* Participation in another clinical trial (use of investigational product or device)
* Not on optimal treatment (COPD patients only)
* Current smokers, exhaled CO >10 parts per million
* Clinical instability, defined as experiencing a COPD exacerbation less than 4 weeks prior to baseline visit, as indicated by treatment with systemic glucocorticosteroids and/or antibiotics and/or hospitalization (COPD only)
* An upper/lower respiratory tract infection e.g. common cold, sinus symptoms, pneumonia, which has not resolved four weeks prior to baseline visit
* Diagnosis of asthma and/or other relevant lung disease (e.g. history of primary or clinically significant bronchiectases, cystic fibrosis, bronchiolitis, lung resection, lung cancer, interstitial lung disease [e.g. fibrosis, silicosis, sarcoidosis], active tuberculosis)
* Known alpha-1-antitrypsin deficiency
* Immunological diseases or known infection with Human Immunodeficiency Virus (HIV)
* Any diagnosis of a malignant disease (other than basal or squamous cell carcinoma) in the last 5 years
* Currently taking immunosuppressive medications
* Diagnosis of diabetes mellitus
* Severe renal failure (calculated eGFR less than 60 ml/min)
* Liver impairment Child-Pugh B/C and/or active viral hepatitis
* Severe psychiatric or neurological disorders (Parkinson's disease or motor neurone disease)
* Planned donation of human tissue (blood, organs or bone marrow) during the course of the trial

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients aged 65-85 years with a diagnosis of COPD (according to Global Initiative for Chronic Obstructive Lung Disease criteria: post bronchodilator FEV1/FVC ratio <0.70) and moderate to severe airflow limitation (FEV1 30-80% predicted) will be approached.
  We will also include healthy participants as a control reference group who are aged 65-85 years without symptoms of lung disease and have normal spirometry.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2016-10; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Haemagglutination inhibition (HI) antibody titres | October 2016 - August 2017

SECONDARY OUTCOMES:
Pseudotype-based neutralization antibody titres | October 2016 - August 2017
Serum and saliva concentrations of total (and sub-classes of) IgA, IgG and IgM | October 2016 - August 2017
Concentrations of inflammatory mediators in RNA extracted from unstimulated and in vitro stimulated peripheral blood mononuclear cells. | October 2016 - August 2017
Plasma concentrations of markers of B and T cell activation | October 2016 - August 2017

CONTACTS AND LOCATIONS:
Overall Officials: Glen Davison, PhD, Principal Investigator — University of Kent
Locations (2):
- United Kingdom (2):
  - Lincolnshire West CCG, Lincoln
  - South Lincolnshire CCG, Lincoln

IPD SHARING:
Plan to Share IPD: No